CLINICAL TRIAL: NCT04492995
Title: Sentinel Node in Endometrial Cancer by Detection of Hybrid ([99mTc] Tc-albumin Nanocoloid-ICG). A Comparative Pilot Study Between the Lymphatic Map Derived From the Cervical Puncture Versus Myometrial
Brief Title: Sentinel Node in Endometrial Cancer
Acronym: HYBRIDENDONOD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Judit Pich Martínez (Other)
Responsible Party: Sponsor-Investigator, Judit Pich Martínez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HYBRID-ENDONODE; 2020-001970-31 (EudraCT Number)
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotracer + TUMIR (Active Comparator): TUMIR = transvaginal ultrsound-guided myometrial injection
  Interventions: Diagnostic Test: injection via TUMIR of the tracer [99mTc] Tc-albumin nanocoloid-ICG (6 mCi, 4 ml)
- (Radiotraces + ICG) + TUMIR (Experimental): ICG =indocyanine green TUMIR = transvaginal ultrsound-guided myometrial injection
  Interventions: Diagnostic Test: injection via TUMIR of [99mTc] Tc-albumin nanocoloid (6mCi, 8ml).

INTERVENTIONS:
Diagnostic Test: injection via TUMIR of the tracer [99mTc] Tc-albumin nanocoloid-ICG (6 mCi, 4 ml) — The day before the surgery, a new scan (planar and SPECT / CT) will be performed after the injection via TUMIR of the tracer [99mTc] Tc-albumin nanocoloid-ICG (6 mCi, 4 ml) or the injection via TUMIR of [99mTc] Tc-albumin nanocoloid (6mCi, 8ml).
  The two lymphatic maps will be compared and the number of sentinel nodes identified in each study and the territories of drainage and the difference between them (in number and territories) will be established.
  On the day of surgery, a cervical injection of methylene blue will be performed at the start of surgery according to usual methodology (2 ml diluted to 50%). Intraoperative detection of the sentinel nodes will take place by visual inspection, using the gammadetector probe and NIR optics. Sentinel node biopsies will be processed according to the usual processing methodology and analysis for the detection of metastases.
  Arms: Radiotracer + TUMIR
Diagnostic Test: injection via TUMIR of [99mTc] Tc-albumin nanocoloid (6mCi, 8ml). — The day before the surgery, a new scan (planar and SPECT / CT) will be performed after the injection via TUMIR of the tracer [99mTc] Tc-albumin nanocoloid-ICG (6 mCi, 4 ml) or the injection via TUMIR of [99mTc] Tc-albumin nanocoloid (6mCi, 8ml).
  The two lymphatic maps will be compared and the number of sentinel nodes identified in each study and the territories of drainage and the difference between them (in number and territories) will be established.
  On the day of surgery, a cervical injection of methylene blue will be performed at the start of surgery according to usual methodology (2 ml diluted to 50%). Intraoperative detection of the sentinel nodes will take place by visual inspection, using the gammadetector probe and NIR optics. Sentinel node biopsies will be processed according to the usual processing methodology and analysis for the detection of metastases.
  Arms: (Radiotraces + ICG) + TUMIR

SUMMARY:
Phase II, open-label, randomized pilot study.

Patients will be randomized (1:1) to receive for sentinel node screening:

1. Radiotracer (RT) via cervical administration and TUMIR
2. Combination of RT with Indocyanine Green (RT + ICG) via cervical administration and TUMIR Patients will be followed up to 1 month after the last administration of radiotracer 70 patients will be included into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histological diagnosis of endometrial cancer with criteria of high risk according to the following criteria: - unfavorable histology according to FIGO (adenocarcinoma serous, clear cell, or carcinosarcoma) - nuclear grade 3 - suspected myometrial invasion> 50% by resonance magnetic (MR) or transvaginal ultrasound
3. Women of childbearing age should have a transvaginal ultrasound who rule out pregnancy and must commit to using methods highly effective contraceptives (vasectomized couple and sexual abstinence) until the hysterectomy is performed.
4. Patient who gives written informed consent.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Suspected lymph node or distant metastatic disease in the preoperative study.
3. History of previous surgery or radiotherapy in the pelvic and paraortic lymphatic drainage areas or nodal involvement of any other etiology.
4. Body mass index (BMI) greater than 45 Kg / m2.
5. Patients who, in the researcher's opinion, are not suitable for participate, regardless of reason, including medical or clinical, or participants potentially at risk of not comply with the study procedures.
6. Known hypersensitivity to some of the active substances or excipients from RT or ICG (including previous history of hypersensitivity to products containing human albumin).
7. Hypersensitivity to sodium iodide.
8. Patients allergic to iodine.
9. Patients with clinical hyperthyroidism, thyroid adenomas autonomic and diffuse focal and autonomic disturbances of the gland thyroid.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with intraoperative detection of sentinel nodes | 1 month

SECONDARY OUTCOMES:
Number of sentinel nodes biopsied during surgery after injection of the [99mTc] hybrid radiotracer Tc-albumin nanocoloid-ICG (hybrid RT) or albumin nanocoloid (RT) radiotracer [99mTc] by myometrial injection guided by transvaginal ultrasound (TUMIR). | 1 month
Number of sentinel lymph nodes with lymph node infiltration detected during surgery after injection of hybrid RT or RT by guided myometrial injection by transvaginal ultrasound (TUMIR) | 1 month
Number of lymph nodes with lymph node infiltration detected in the piece of lymphadenectomy after injection of hybrid RT or RT by TUMIR injection lymphadenectomy after injection of hybrid RT or RT by TUMIR injection | 1 month
Number of false negative results after injection of the hybrid RT or RT by transvaginal ultrasound-guided myometrial injection (TUMIR). | 1 month
Difference in the number of sentinel nodes visualized after injection of the hybrid RT or RT between TUMIR lymphogammagraphy and cervical lymphogammagraphy | 1 month
Difference in the drainage pattern of each radiotracer (hybrid RT and RT) between the cervical injection and transvaginal ultrasound-guided myometrial injection (TUMIR). | 1 month
Causes of non-drainage of the hybrid RT or RT in the cervical injection or in the Transvaginal ultrasound-guided myometrial injection (TUMIR). | 1 month
Difference between the proportion of paraortic sentinel nodes detected after injection of each of the radiotracers (hybrid RT and RT) during surgery. | 1 month
Proportion of patients with hypersensitivity reactions related to injection of each of the two radiotracers (hybrid RT and RT). | 1 month
Proportion of patients with adverse events related to injection of one of the two radiotracers (hybrid RT and RT). | 1 month
Surgical detection time of sentinel nodes during intraoperative detection after injection of each of the two radiotracers (hybrid RT and RT). | 1 month
Histological data of the tumor: histology, tumor grade, tumor size and myometrial infiltration. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Paredes, MD, Principal Investigator — Hospital Clinic of Barcelona; Sergi Vidal, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] van Oosterom MN, Diaz-Feijoo B, Santisteban MI, Sanchez-Izquierdo N, Perissinotti A, Glickman A, Marina T, Torne A, van Leeuwen FWB, Vidal-Sicart S. Steerable DROP-IN radioguidance during minimal-invasive non-robotic cervical and endometrial sentinel lymph node surgery. Eur J Nucl Med Mol Imaging. 2024 Aug;51(10):3089-3097. doi: 10.1007/s00259-023-06589-3. Epub 2024 Jan 18. PMID 38233608